CLINICAL TRIAL: NCT04626479
Title: A Phase 1b/2 Study of Immune and Targeted Combination Therapies in Participants With RCC (U03): Substudy 03A in First Line Metastatic Participants
Brief Title: Substudy 03A: A Study of Immune and Targeted Combination Therapies in Participants With First Line (1L) Renal Cell Carcinoma (MK-3475-03A)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-03A; MK-3475-03A (Other: MSD); 2023-506838-68-00 (Registry Identifier: EU CT); U1111-1294-4527 (Registry Identifier: UTN); 2019-003609-84 (EudraCT Number)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: receptor tyrosine kinase inhibitor; programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; belzutifan; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Coformulation Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants will receive pembrolizumab/quavonlimab (coformulation of pembrolizumab 400 mg and quavonlimab 25 mg) PLUS lenvatinib 20 mg. Pembrolizumab/quavonlimab will be administered intravenously (IV) once every 6 weeks (Q6W) for up to 17 administrations (up to ~2 years). Lenvatinib will be administered orally once-daily (QD) until progressive disease or discontinuation.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab/Quavonlimab
- Coformulation Favezelimab/Pembrolizumab+ Lenvatinib (Experimental): Participants will receive favezelimab/pembrolizumab (coformulation of favezelimab 800 mg and pembrolizumab 200 mg) PLUS lenvatinib 20 mg. Favezelimab/Pembrolizumab will be administered IV once every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Favezelimab/Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab + Belzutifan + Lenvatinib (Experimental): Participants will receive pembrolizumab 400 mg PLUS belzutifan 120 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered IV Q6W for up to 17 administrations (up to ~2 years). Both belzutifan and lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Belzutifan; Drug: Lenvatinib
- Pembrolizumab + Lenvatinib (Experimental): Participants will receive pembrolizumab 400 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered IV Q6W for up to 17 administrations (up to ~ 2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Coformulation Vibostolimab/Pembrolizumab+Belzutifan (Experimental): Participants will receive vibostolimab/pembrolizumab (coformulation of 200 mg vibostolimab and pembrolizumab 200 mg). Vibostolimab/pembrolizumab will be administered IV once every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years). Belzutifan will be administered orally QD until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Vibostolimab/Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered via IV infusion at a dose of 400 mg Q6W
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Belzutifan + Lenvatinib; Pembrolizumab + Lenvatinib
Biological: Favezelimab/Pembrolizumab — Administered via IV infusion at a dose of 800 mg/200 mg Q3W
  Other Names: MK-4280A
  Arms: Coformulation Favezelimab/Pembrolizumab+ Lenvatinib
Drug: Belzutifan — Administered via oral tablet at a dose of 120 mg QD
  Other Names: MK-6482; WELIREG™
  Arms: Coformulation Vibostolimab/Pembrolizumab+Belzutifan; Pembrolizumab + Belzutifan + Lenvatinib
Drug: Lenvatinib — Administered via oral capsule at a dose of 20 mg QD
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Coformulation Favezelimab/Pembrolizumab+ Lenvatinib; Coformulation Pembrolizumab/Quavonlimab + Lenvatinib; Pembrolizumab + Belzutifan + Lenvatinib; Pembrolizumab + Lenvatinib
Biological: Pembrolizumab/Quavonlimab — Administered via IV infusion at a dose of 400 mg/25 mg Q6W
  Other Names: MK-1308A
  Arms: Coformulation Pembrolizumab/Quavonlimab + Lenvatinib
Drug: Vibostolimab/Pembrolizumab — Administered via IV infusion at a dose of 200 mg/200 mg Q6W
  Other Names: MK-7684A
  Arms: Coformulation Vibostolimab/Pembrolizumab+Belzutifan

SUMMARY:
Substudy 03A is part of a larger research study that is testing experimental treatments for renal cell carcinoma (RCC). The larger study is the umbrella study (U03).

The goal of substudy 03A is to evaluate the safety and efficacy of experimental combinations of investigational agents in participants with advanced first line (1L) clear cell renal cell carcinoma (ccRCC).

This substudy will have two phases: a safety lead-in phase and an efficacy phase. The safety lead-in phase will be used to demonstrate a tolerable safety profile for the combination of investigational agents. There will be no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of locally advanced/metastatic ccRCC
* Has received no prior systemic therapy for advanced RCC; prior neoadjuvant/adjuvant therapy for RCC is acceptable if completed ≥12 months before randomization/allocation.
* Is able to swallow oral medication
* Has adequate organ function
* Participants receiving bone resorptive therapy must have therapy initiated at least 2 weeks before randomization/allocation
* Has resolution of toxic effects of the most recent prior therapy to ≤Grade 1
* Has adequately controlled blood pressure (BP ≤150/90 mm Hg) with no change in hypertensive medications within 1 week before randomization/allocation
* Male participants are abstinent from heterosexual intercourse or agree to use contraception during treatment with and for at least 7 days after the last dose of lenvatinib and /or belzutifan; 7 days after lenvatinib and/or belzutifan is stopped, if the participant is only receiving pembrolizumab, pembrolizumab/quavonlimab, favezelimab/pembrolizumab or a combination of the aforementioned drugs, no contraception is needed
* Female participants must not be pregnant and not be a woman of childbearing potential (WOCBP) or is a WOCBP abstinent from heterosexual intercourse or using contraception during the intervention period and for at least 120 days after the last dose of pembrolizumab, pembrolizumab/quavonlimab, favezelimab/pembrolizumab for 30 days after the last dose of lenvatinib or belzutifan, whichever occurs last and must abstain from breastfeeding during the study intervention period and for at least 120 days after study intervention

Exclusion Criteria:

* Has urine protein ≥1 g/24 hours and has any of the following: (a) a pulse oximeter reading <92% at rest, or (b) requires intermittent supplemental oxygen, or (c) requires chronic supplemental oxygen (d) active hemoptysis within 3 weeks prior to the first dose of study intervention
* Has clinically significant cardiovascular disease within 12 months from the first dose of study intervention administration
* Has had major surgery within 3 weeks before first dose of study interventions
* Has a history of lung disease
* Has a history of inflammatory bowel disease
* Has preexisting gastrointestinal (GI) or non-GI fistula
* Has malabsorption due to prior GI surgery or disease
* Has received prior radiotherapy within 2 weeks of start of study intervention
* Has received a live or live attenuated vaccine within 30 days before the first dose of study drug; killed vaccines are allowed
* Has received more than 4 previous systemic anticancer treatment regimens
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years; replacement therapy is not considered a form of systemic treatment and is allowed
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B
* Has had an allogenic tissue/solid organ transplant

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Phase: Number of participants who experience one or more dose-limiting toxicities (DLTs) | Up to ~21 days
  DLTs are defined as one or more of the following toxicities: (1) grade (gr) 4 nonhematologic toxicity (2) gr 4 hematologic toxicity lasting >7 days OR gr 4 platelet count decreased of any duration OR gr 3 platelet count decreased if associated with bleeding (3) gr 3 nonhematologic toxicity except gr 3 fatigue (lasting ≤3 days), diarrhea, nausea, vomiting or rash without standard of care (4) gr 3 or 4 nonhematologic abnormality if medical intervention is required or if it leads to hospitalization or persists for >1 week (5) gr 3 or 4 febrile neutropenia (6) gr 3 or 4 alanine aminotransferase, aspartate aminotransferase and/or bilirubin laboratory value (7) treatment related adverse event (AE) causing study intervention discontinuation during the first 21 days (8) treatment related AE causing intervention administration delay for >14 days during the first 21 days (9) gr 5 toxicity. The number of participants who experience one or more DLTs in the safety lead-in phase will be presented.
Safety Lead-in Phase: Number of participants who experience one or more adverse events (AEs) | Up to ~21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs in the safety lead-in phase will be presented.
Safety Lead-in Phase: Number of participants who discontinue study treatment due to an AE | Up to ~21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE in the safety lead-in phase will be presented.
Efficacy Phase: Number of participants who experience one or more DLTs | Up to ~21 days
  DLTs are defined as one or more of the following toxicities: (1) grade (gr) 4 nonhematologic toxicity (2) gr 4 hematologic toxicity lasting >7 days OR gr 4 platelet count decreased of any duration OR gr 3 platelet count decreased if associated with bleeding (3) gr 3 nonhematologic toxicity except gr 3 fatigue (lasting ≤3 days), diarrhea, nausea, vomiting or rash without standard of care (4) gr 3 or 4 nonhematologic abnormality if medical intervention is required or if it leads to hospitalization or persists for >1 week (5) gr 3 or 4 febrile neutropenia (6) gr 3 or 4 alanine aminotransferase, aspartate aminotransferase and/or bilirubin laboratory value (7) treatment related adverse event (AE) causing study intervention discontinuation during the first 21 days (8) treatment related AE causing intervention administration delay for >14 days during the first 21 days (9) gr 5 toxicity. The number of participants who experience one or more DLTs in the efficacy phase will be presented.
Efficacy Phase: Number of participants who experience one or more AEs | Up to ~43 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs in the efficacy phase will be presented.
Efficacy Phase: Number of participants who discontinue study treatment due to an AE | Up to ~43 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE in the efficacy phase will be presented.
Efficacy Phase: Objective response rate (ORR) | Up to ~43 months
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Efficacy Phase: Duration of response (DOR) | Up to ~43 months
  For participants in the analysis population who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters), DOR is defined as the time from first documented evidence of CR or PR until progressive disease or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 by BICR.
Efficacy Phase: Progression-free survival (PFS) | Up to ~43 months
  PFS is defined as the time from randomization to the first documented progressive disease or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 by BICR.
Efficacy Phase: Overall survival (OS) | Up to ~43 months
  OS is defined as the time from randomization to death due to any cause.
Efficacy Phase: Clinical benefit rate (CBR) | Up to ~43 months
  CBR is defined as the percentage of participants who have achieved CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) of ≥6 months. Responses are according to RECIST 1.1 by BICR.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (55):
- United States (10):
  - University of California at San Francisco ( Site 1008), San Francisco, California
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 1011), New Haven, Connecticut
  - University of Chicago ( Site 1013), Chicago, Illinois
  - University of Iowa ( Site 1012), Iowa City, Iowa
  - Henry Ford Health System ( Site 1014), Detroit, Michigan
  - Laura and Isaac Perlmutter Cancer Center ( Site 1016), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1002), New York, New York
  - Duke Cancer Institute ( Site 1015), Durham, North Carolina
  - UPMC Cancer Center/Hillman Cancer Center ( Site 1017), Pittsburgh, Pennsylvania
  - UTSW Medical Center ( Site 1003), Dallas, Texas
- Australia (4):
  - Western Sydney Local Health District ( Site 1601), Blacktown, New South Wales
  - St George Hospital ( Site 1602), Kogarah, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 1603), Herston, Queensland
  - Austin Health ( Site 1600), Heidelberg, Victoria
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 1101), Toronto, Ontario
  - Jewish General Hospital ( Site 1100), Montreal, Quebec
- Chile (6):
  - FALP-UIDO ( Site 2100), Santiago, Region M. de Santiago
  - Oncovida ( Site 2107), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 2101), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 2108), Temuco, Región de la Araucanía
  - CIDO SpA-Oncology ( Site 2106), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 2103), Viña del Mar, Región de Valparaíso
- Colombia (4):
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 1900), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 1905), Valledupar, Cesar Department
  - Oncomédica S.A.S ( Site 1904), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 1901), Cali, Valle del Cauca Department
- France (4):
  - Institut De Cancerologie De Lorraine ( Site 1204), Vandœuvre-lès-Nancy, Ain
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 1203), Strasbourg, Alsace
  - Institut Claudius Regaud ( Site 1200), Toulouse, Haute-Garonne
  - Gustave Roussy ( Site 1202), Villejuif, Val-de-Marne
- Országos Onkológiai Intézet-Urogenitális Tumorok és Klinikai Farmakológiai Osztály ( Site 2301), Budapest, Pest County, Hungary
- Israel (5):
  - Rambam MC ( Site 1500), Haifa
  - Hadassah Medical Center-Oncology ( Site 1504), Jerusalem
  - Rabin Medical Center ( Site 1502), Petah Tikva
  - Sheba Medical Center - Oncology Division ( Site 1501), Ramat Gan
  - Sourasky Medical Center ( Site 1503), Tel Aviv
- Netherlands (2):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL)-medical oncology ( Site 2402), Amsterdam, North Holland
  - Erasmus Medisch Centrum ( Site 2401), Rotterdam, South Holland
- Auckland City Hospital ( Site 1700), Auckland, New Zealand
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2201), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 2200, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 2202), Gdansk, Pomeranian Voivodeship
- South Korea (3):
  - Asan Medical Center ( Site 1800), Songpagu, Seoul
  - Severance Hospital ( Site 1802), Seoul
  - Samsung Medical Center ( Site 1801), Seoul
- Spain (2):
  - Hospital Universitari Vall d Hebron ( Site 1300), Barcelona, Catalonia
  - Hospital Universitario Ramon y Cajal ( Site 1301), Madrid
- United Kingdom (8):
  - Southampton General Hospital ( Site 1403), Southampton, England
  - The Beatson West of Scotland Cancer Centre ( Site 1405), Glasgow, Glasgow City
  - Royal Preston Hospital ( Site 1406), Preston, Lancashire
  - Leicester Royal Infirmary ( Site 1408), Leicester, Leicestershire
  - Barts Health NHS Trust ( Site 1401), London, London, City of
  - Western General Hospital ( Site 1402), Edinburgh, Midlothian
  - Velindre Cancer Centre Hospital ( Site 1407), Cardiff, Wales
  - The Christie NHS Foundation Trust ( Site 1400), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Suarez C, Rojas C, Shin SJ, Yanez Weber P, Albiges L, Motzer R, Hammers H, Peer A, Lee JL, Miller WH, Waddell T, Neiman V, Keizman D, Zwenger Kloster A, Weickhardt A, Dziadziuszko R, Suttner L, Sharma M, Burgents JE, Powles T. Novel pembrolizumab-based treatments as first-line therapy in advanced clear-cell renal cell carcinoma: substudy 03A of the open-label, umbrella platform, phase I/II KEYMAKER-U03 trial. Ann Oncol. 2026 Feb;37(2):229-240. doi: 10.1016/j.annonc.2025.10.010. Epub 2025 Oct 18. PMID 41115468
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26225&tenant=MT_MSD_9011